CLINICAL TRIAL: NCT03730870
Title: Assessment of Pharmacogenomics Testing for Improving Pediatric ADHD Psychopharmacological Treatment: A Randomized Controlled Trial
Brief Title: Pharmacogenomics for Improving Pediatric ADHD Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study's genetic testing laboratory has suspended operations pending discussions with the FDA concerning clinical interpretation of pharmacogenomics tests.
Sponsor: Clinical and Translational Genome Research Institute, Inc. (Other)
Collaborators: Children's Specialized Hospital (Other)
Responsible Party: Principal Investigator, Dan Handley, M.S., Ph.D., Chief Scientific Officer, Clinical and Translational Genome Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-01
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Attention Deficit Disorders With Hyperactivity
Keywords: Attention Deficit Disorders with Hyperactivity; ADHD; Pharmacogenomics; Pediatric ADHD; ADHD medications
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to have their study clinician have access to their pharmacogenomics report prior to prescribing medications (experimental group) or no access (control group) until end of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinded as to study arm participation and outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pharmacogenomics report (Experimental): Clinician reviews pharmacogenomics report for subject prior to prescribing FDA-approved medications.
  Interventions: Diagnostic Test: Pharmacogenomics report
- Control (No Intervention): Clinician prescribes FDA-approved medications as customarily performed without additional guidance from pharmacogenomics report ("treatment-as-usual").

INTERVENTIONS:
Diagnostic Test: Pharmacogenomics report — Intervention is the performance of a pharmacogenomics laboratory-developed test (LDT) performed by high-throughput sequencing of 38 genes involved in drug pharmacokinetics or pharmacodynamics. The clinician reviews the report results for each subject.
  Arms: Pharmacogenomics report

SUMMARY:
This research study is a randomized controlled trial (RCT) to test whether pharmacogenomics (PGx) testing for ADHD medications will help guide clinicians to choose medications and dosages for pediatric ADHD treatment that provide faster symptom relief, fewer or less severe side effects, improve patient quality of life, and lessen emotional stress for parents/guardians of the patients.

DETAILED DESCRIPTION:
The study is a randomized controlled trial (RCT) of pediatric Attention Deficit Hyperactivity Disorder (ADHD) patients using an experimental group and a control group. The subjects in the experimental group will be administered a commercially available pharmacogenomics (PGx) test panel of 38 genes specifically related to drug metabolism rates and drug response. A subset of these genes are known to be involved in the pharmacokinetics and pharmacodynamics of ADHD medications.

The PGx test report indicates if there are genetic variants detected related to ADHD medications and consequently provides recommendations for the clinician on which medications and doses may be optimally effective. The control group is the "treatment as usual" (TAU) group whose subjects are treated with medications for ADHD based on the treating clinician's customary method(s) for selecting medications and doses.

The hypotheses to be tested are that PGx testing guidance will reduce the time it takes to reach a treatment regimen that improves patient symptom relief, reduces the frequency and severity of adverse drug reactions, improves patient quality of life, and reduces parental emotional stress. Additionally, since the test is performed using next-generation sequencing, we wish to tabulate relevant allele frequencies and use variant call files to discover previously unknown PGx genetic variants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 6 and 18 inclusive at the start of the study.
* Provision of signed and dated informed consent form.
* Subject and parent or legal guardian must state willingness to comply with all study procedures and availability for the duration of the study.
* Both male and female subjects will be recruited from the pediatric population diagnosed with any subtype of ADHD without Oppositional Defiant Disorder (ODD) via the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria.
* Subject and their parent or legal guardian will read and speak English with sufficient proficiency to understand the study and be able to give informed assent and consent.
* Subject will be able to complete study procedures such as filling out paper quality of life assessments
* Subjects will be able to take oral medication(s) if and as prescribed.
* Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

* Subjects will not have been treated for any condition with psychiatric prescription medications within the previous six (6) months.
* Subjects will not have had a diagnosis of Oppositional Defiant Disorder (ODD).
* Subject will not be currently a suicide risk, has previously made a suicide attempt or has a prior history of suicidal behavior.
* Subject will not have a history of alcohol or other substance abuse or dependence within the last 6 months.
* Subject will not have used an investigational medicinal product or participation in a clinical study within six (6) months prior to the baseline visit.
* Subject will not have a clinically important abnormality on urine drug and alcohol screen, if one had been taken.
* If the subject is female, is not currently pregnant, reasonably expecting to become pregnant, or lactating.
* Subject will not have a known or suspected allergy to any of the potential medications that may be prescribed.
* Only one subject per family will be enrolled to prevent systematic bias based on a parent or legal guardian's personal style of symptom assessment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Assessment of Change in ADHD Symptom Severity Between Experimental and Control Group | At baseline and at 24 weeks
  Measurement is performed by using the National Institute for Children's Health Quality (NICHQ) Vanderbilt Assessment Scales. The Vanderbilt assessment for ADHD is a validated questionnaire that provides a quantitative measure of ADHD symptoms and severity. Specific measures:
  Symptom Score: 18 questions on symptom type and severity between a measure of 0 (Never) and 3 (Very Often). Total Symptom Score range from 0 to 54. Lower scores indicate less severe symptoms.
  Performance Score: 8 questions on subject academic and interpersonal relationship functions using a measure between 1 (Excellent) and 5 (Problematic). Performance Score ranges from 0 to 40. Lower scores indicate better performance.
  Side Effects or Problems: 12 questions related to health and behavioral issues. Scores range from None, Mild, Moderate, to Severe. These are not quantitatively scored on the assessment.
  These measurements will be analyzed separately.
  This assessment is performed by parent/guardian.

SECONDARY OUTCOMES:
Assessment of Differences in Parenting Stress Between Experimental and Control Group | At baseline and at 24 weeks
  Measurement is performed using the Psychological Assessment Resources (PAR) Parenting Stress Index - 4th edition - Short Form for Parents of Children (ages 6-10) or Stress Index for Parents of Adolescents (ages 11-18) as appropriate for age at time of enrollment.
  Questionnaire for children ages 6 - 10 consists of 36 questions regarding problems with parental stress. Scale for each question ranges from 1 (Strongly Agree) to 5 (Strongly Disagree). Total scoring ranges from 36 to 180. Higher scores indicate less parenting stress.
  Questionnaire for adolescents ages 11 - 18 consists of 90 questions regarding problems with parental stress. Scale for each question ranges from 1 (Strongly Agree) to 5 (Strongly Disagree). Total scoring ranges from 90 to 450. Higher scores indicate less parenting stress.
  Assessment performed by parent/guardian.
Assessment of Differences in Child's Quality of Life Between Experimental and Control Group | At baseline and at 24 weeks
  Measurement is performed using the PedsQL Pediatric Quality of Life Inventory Parent-Proxy Report for Children (ages 5-7, 8-12, 13-18).
  Questionnaire consists of 23 questions regarding problems with subject's physical, emotional, social, and school functioning. Scale for each question ranges from 0 (Never) to 4 (Almost Always). Total scoring ranges from 0 to 92. Lower scores indicate higher quality of life.
  Assessment is performed by parent/guardian.
Self-assessment of Differences in Child's Quality of Life Between Experimental and Control Group | At baseline and at 24 weeks
  Measurement is performed using the PedsQL Pediatric Quality of Life Inventory Child-Self Report (ages 5-7, 8-12, 13-18).
  Questionnaire consists of 23 questions regarding problems with subject's physical, emotional, social, and school functioning. Scale for each question ranges from 0 (Never) to 4 (Almost Always). Total scoring ranges from 0 to 92. Lower scores indicate higher quality of life.
  Assessment performed by subject.

OTHER OUTCOMES:
PGx Allele Frequency Tabulation | 1 year from start of study
  Tabulation of allele frequencies associated with the PGx genes that are sequenced. This is intended to add to current knowledge of how prevalent relevant alleles are in the population.
Analysis of variant call files for genetic variants | 1 year from start of study
  Analysis of next-generation sequencing variant call files to determine whether the tests capture any previously unknown or undiscovered genetic variants, and assess their possible clinical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Handley, M.S., Ph.D., Principal Investigator — Clinical and Translational Genome Research Institute, Inc.
Locations (3):
- United States (3):
  - Children's Specialized Hospital, Hamilton, New Jersey
  - Children's Specialized Hospital, Mountainside, New Jersey
  - Children's Specialized Hospital, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Botkin JR, Belmont JW, Berg JS, Berkman BE, Bombard Y, Holm IA, Levy HP, Ormond KE, Saal HM, Spinner NB, Wilfond BS, McInerney JD. Points to Consider: Ethical, Legal, and Psychosocial Implications of Genetic Testing in Children and Adolescents. Am J Hum Genet. 2015 Jul 2;97(1):6-21. doi: 10.1016/j.ajhg.2015.05.022. PMID 26140447
- [Background] Smith T, Sharp S, Manzardo AM, Butler MG. Pharmacogenetics informed decision making in adolescent psychiatric treatment: a clinical case report. Int J Mol Sci. 2015 Feb 20;16(3):4416-28. doi: 10.3390/ijms16034416. PMID 25710722
- [Background] Olson MC, Maciel A, Gariepy JF, Cullors A, Saldivar JS, Taylor D, Centeno J, Garces JA, Vaishnavi S. Clinical Impact of Pharmacogenetic-Guided Treatment for Patients Exhibiting Neuropsychiatric Disorders: A Randomized Controlled Trial. Prim Care Companion CNS Disord. 2017 Mar 16;19(2). doi: 10.4088/PCC.16m02036. PMID 28314093
- [Background] Gomez-Sanchez CI, Carballo JJ, Riveiro-Alvarez R, Soto-Insuga V, Rodrigo M, Mahillo-Fernandez I, Abad-Santos F, Dal-Re R, Ayuso C. Pharmacogenetics of methylphenidate in childhood attention-deficit/hyperactivity disorder: long-term effects. Sci Rep. 2017 Sep 4;7(1):10391. doi: 10.1038/s41598-017-10912-y. PMID 28871191
- [Background] Polanczyk G, Zeni C, Genro JP, Roman T, Hutz MH, Rohde LA. Attention-deficit/hyperactivity disorder: advancing on pharmacogenomics. Pharmacogenomics. 2005 Apr;6(3):225-34. doi: 10.1517/14622416.6.3.225. PMID 16013954
- [Background] Myer NM, Boland JR, Faraone SV. Pharmacogenetics predictors of methylphenidate efficacy in childhood ADHD. Mol Psychiatry. 2018 Sep;23(9):1929-1936. doi: 10.1038/mp.2017.234. Epub 2017 Dec 12. PMID 29230023
- [Background] Wehry AM, Ramsey L, Dulemba SE, Mossman SA, Strawn JR. Pharmacogenomic Testing in Child and Adolescent Psychiatry: An Evidence-Based Review. Curr Probl Pediatr Adolesc Health Care. 2018 Feb;48(2):40-49. doi: 10.1016/j.cppeds.2017.12.003. Epub 2018 Jan 8. PMID 29325731